CLINICAL TRIAL: NCT01123967
Title: Improved Effectiveness of Smoking Cessation Programs for Minnesota Priority Populations
Brief Title: Offering Proactive Tobacco Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2009NTLS064; 0909S72235 (Other: IRB, University of Minnesota); 1R01CA141527 (NIH)
Record Dates: First submitted 2010-05-12; First posted 2010-05-14 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Tobacco Use Cessation
Keywords: nicotine replacement therapy; smoking cessation; tobacco dependent
MeSH Terms: conditions — Tobacco Use Cessation; Smoking Cessation | interventions — Nicotine Replacement Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PRO+NRT+TC (Experimental): Proactive outreach (mailed invitation letter followed by telephone outreach) combined with free nicotine replacement therapy (NRT) and telephone counseling (PRO+NRT+TC)to usual care (UC)
  Interventions: Other: proactive outreach (PRO); Other: telephone counseling (TC); Other: Nicotine replacement therapy (NRT)
- Usual Care (UC) (Active Comparator): Usual (standard) care - Smoking cessation products: patch, gum, lozenge, inhaler and nasal spray
  Interventions: Other: Usual care (UC)

INTERVENTIONS:
Other: proactive outreach (PRO) — a mailed invitation letter followed by telephone outreach
  Arms: PRO+NRT+TC
Other: telephone counseling (TC) — free telephone counseling
  Arms: PRO+NRT+TC
Other: Nicotine replacement therapy (NRT) — free nicotine replacement therapy (NRT)
  Arms: PRO+NRT+TC
Other: Usual care (UC) — nicotine replacement products (patch, gum, lozenge, inhaler, and nasal spray)
  Arms: Usual Care (UC)

SUMMARY:
This study uses a proactive outreach strategy, coupled with free nicotine replacement therapy (NRT) to increase the population impact of tobacco cessation treatment for diverse, low income smokers. Population impact is the product of treatment utilization (i.e., reach or exposure) and treatment efficacy (i.e., smoking abstinence rates among those who utilize treatment).

DETAILED DESCRIPTION:
Participants will be randomized to receive either Usual (Reactive) Care or Proactive Outreach, Telephone Counseling and free nicotine replacement therapy (NRT).

ELIGIBILITY:
Inclusion Criteria:

* Must complete the baseline survey
* Current self-reported cigarette smoker
* Has a valid home address
* An adequate proficiency in English to complete study surveys and participate in telephone counseling.

exclusion Criteria:

* adult smokers not enrolled in the Minnesota Health Care Programs (MHCP).

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2500 (Actual)
Dates: Start 2011-02; Primary Completion 2014-02 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Results in Abstinence Rates | 1 Year
  Compare the effect of proactive outreach combined with free NRT and telephone counseling (PRO+NRT+TC) to usual care (UC) on population-level smoking abstinence rates among a diverse population of low income smokers.

SECONDARY OUTCOMES:
Results in Treatment Utilization | 1 Year
  Compare the effect of proactive outreach combined with free NRT and telephone counseling (PRO+NRT+TC) to usual care (UC) on population-level tobacco treatment utilization rates among a diverse population of low income smokers.
Cost-Effectiveness of Program | 1 Year
  Determine the cost-effectiveness of PRO+NRT+TC compared with UC.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Fu, M.D., Principal Investigator — Veterans Administration Hospital; Anne Joseph, MD, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- Steven Fu, M.D., Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Hammett PJ, Japuntich SJ, Sherman SE, Rogers ES, Danan ER, Noorbaloochi S, El-Shahawy O, Burgess DJ, Fu SS. Proactive tobacco treatment for veterans with posttraumatic stress disorder. Psychol Trauma. 2021 Jan;13(1):114-122. doi: 10.1037/tra0000613. Epub 2020 Jul 2. PMID 32614201
- [Derived] Hammett PJ, Lando HA, Erickson DJ, Widome R, Taylor BC, Nelson D, Japuntich SJ, Fu SS. Proactive outreach tobacco treatment for socioeconomically disadvantaged smokers with serious mental illness. J Behav Med. 2020 Jun;43(3):493-502. doi: 10.1007/s10865-019-00083-8. Epub 2019 Jul 30. PMID 31363948
- [Derived] Fu SS, van Ryn M, Nelson D, Burgess DJ, Thomas JL, Saul J, Clothier B, Nyman JA, Hammett P, Joseph AM. Proactive tobacco treatment offering free nicotine replacement therapy and telephone counselling for socioeconomically disadvantaged smokers: a randomised clinical trial. Thorax. 2016 May;71(5):446-53. doi: 10.1136/thoraxjnl-2015-207904. Epub 2016 Mar 1. PMID 26931362
- [Derived] Fu SS, van Ryn M, Burgess DJ, Nelson D, Clothier B, Thomas JL, Nyman JA, Joseph AM. Proactive tobacco treatment for low income smokers: study protocol of a randomized controlled trial. BMC Public Health. 2014 Apr 9;14:337. doi: 10.1186/1471-2458-14-337. PMID 24716466